CLINICAL TRIAL: NCT07360041
Title: Are Extracorporeal Shock Wave Lithotripsy and Mini-Percutaneous Nephrolithotomy Equivalent in The Management of Pediatric High-Density Renal Stones? A Prospective Randomized Study
Brief Title: Comparison of ESWL and Mini-PCNL for High-Density Renal Stones in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASUMD127/2023
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Renal Stones; Calculus; Pediatric; Endoscopy
Keywords: 10-20 mm non lower calyceal high density renal stones; renal; calculus; pediatrics; ESWL; PCNL
MeSH Terms: conditions — Nephrolithiasis; Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Miniaturized Percutaneous Nephrolithotomy (mini-PNL) (Active Comparator): Miniaturized Percutaneous Nephrolithotomy (mini-PNL)
  Interventions: Procedure: Miniaturized Percutaneous Nephrolithotomy (mini-PNL)
- Shock Wave Lithotripsy (SWL) (Active Comparator): Shock Wave Lithotripsy (SWL)
  Interventions: Procedure: Shock Wave Lithotripsy (SWL)

INTERVENTIONS:
Procedure: Miniaturized Percutaneous Nephrolithotomy (mini-PNL) — Mini-PNL: All procedures will be done in the prone position. The target calyx will be punctured using fluoroscopic guidance with an 18-GA sheathed needle, and tract dilatation will be achieved using Amplantz dilators up to 16-18 Fr according to patient age. The holmium: YAG laser will be used to perform the stone fragmentation. Standard 12-Fr rigid nephroscope will be used for stone retrieval and fragmentation. A clamped nephrostomy tube will be placed routinely to reduce the bleeding for 24 h in all cases. The nephrostomy tube and the ureteral catheter will be removed on first and second postoperative days if there will be no complications.
  Arms: Miniaturized Percutaneous Nephrolithotomy (mini-PNL)
Procedure: Shock Wave Lithotripsy (SWL) — The lithotripsy will be performed by an electromagnetic shockwave lithotripter (Dornier Compact Sigma). The lung and genitourinary fields will be shielded for all patients. Fluoroscopy will be used to localize the stone and to monitor fragmentation.The dispensed shockwave will begin at 14 kV and escalates to its maximum power level of 20 kV. The maximum number of shocks given per session will be between 1000 and 2500 depending on patient age (1000 waves per session for children younger than 5 years and 2500 waves per session for older children, with a frequency of 70 shocks/minute). The SWL session will be stopped when no visible stone is detected, or when tiny fragments are the only visible stone remnants, or when the desired number of shocks has been given.
  Arms: Shock Wave Lithotripsy (SWL)

SUMMARY:
Pediatric nephrolithiasis is an increasing health problem, with rising prevalence particularly in certain geographic regions. Management options for pediatric renal stones include extracorporeal shockwave lithotripsy (SWL), percutaneous nephrolithotomy (PNL), and retrograde intrarenal surgery. According to the EAU/ESPU guidelines, SWL is recommended as a first-line treatment for most renal stones; however, its success is significantly influenced by stone size, location, and density. High-density renal stones (≥1000 Hounsfield Units) are associated with lower stone-free rates after SWL and higher retreatment rates.

Miniaturized percutaneous nephrolithotomy (mini-PNL) has emerged as an effective alternative, offering high stone-free rates with reduced morbidity compared to standard PNL due to the use of smaller access sheaths. While adult studies have demonstrated superior outcomes of mini-PNL over SWL for high-density renal stones, there is a lack of comparative data in the pediatric population.

This prospective randomized controlled study aims to compare the efficacy and safety of mini-PNL versus SWL in children aged 2 to 12 years with single, non-lower pole, high-density (≥1000 HU), medium-sized (10-20 mm) renal stones. Eligible patients will be randomized into two equal groups to undergo either mini-PNL or SWL under general anesthesia.

The primary outcome is the stone-free rate, defined as no residual stone or residual fragments ≤4 mm on non-contrast computed tomography performed three months after the procedure. Secondary outcomes include operative and fluoroscopy times, hemoglobin drop, length of hospital stay, retreatment and ancillary procedure rates, and postoperative complications graded according to the Clavien-Dindo classification.

The study will be conducted at a single tertiary referral center. All participants' parents or legal guardians will provide informed consent in accordance with Good Clinical Practice guidelines and the Declaration of Helsinki. This study aims to provide evidence to guide optimal management of pediatric patients with high-density renal stones.

DETAILED DESCRIPTION:
INTRODUCTION:

While nephrolithiasis is far more common in adults, pediatric stone disease is increasing in prevalence, especially in adolescent females , with higher incidences in the Middle East and North Africa and less common in North America and Europe . The management of pediatric upper urinary tract stones includes extracorporeal shockwave lithotripsy (SWL), percutaneous nephrolithotomy (PNL), and retrograde intrarenal surgery (RIRS).

SWL is a non-invasive procedure that can be performed in children. The European Association of Urology and European Society for Pediatric Urology (EAU/ESPU) guidelines recommend SWL as the primary treatment option for majority of renal stones and upper ureter stones. The stone-free rate (SFR) is significantly affected by various factors; stone location, size and density. Also, presence and degree of obstruction/impaction, and stone-to-skin distance affect SFR. SWL has SFR of nearly 90% for stones <1 cm, 80% for 1-2 cm, 60% for >2 cm. Concerns about anaesthesia and high retreatment rate represent SWL drawback .

The EAU/ESPU guidelines recommend PNL as a mainline of treatment in renal stones larger than 2 cm in the renal pelvis or more than 1 cm in lower pole stone as well as staghorn stones , as the SFR of PNL is between 86.9% and 98.5% after a single session, even in complete staghorn cases, it has a clearance rate of 89%. The PNL complications in children include bleeding, postoperative fever or infection, and persistent urinary leakage. With the miniaturised PNL (mini-PNL) through a 16-18F sheath, the transfusion rates and complications decreased.

The EAU/ESPU guidelines recommended SWL as a primary treatment for renal pelvis, 10-20 mm . However, some authors reported that SWL in children was more successful for stones with HU <1000.Also, in another recent study for adult patients with single, non-lower pole, high-density (≥1000 HU) renal stones, the SFR was 97.1% in the mini-PNL group versus 30.3% in the SWL group .

To the best of our knowledge, no studies in the pediatric population compared mini-PNL and SWL for single, non-lower pole, high-density (≥1000 HU) medium sized renal stones. In this study we will try to fill this gap in the literature

AIM OF THE STUDY:

To compare the outcomes of miniaturised percutaneous nephrolithotomy (mini-PNL) and extracorporeal shockwave lithotripsy (SWL) in the management of 10-20 mm, non-lower pole, high-density (≥1000 HU) renal stones in the pediatric population.

PATIENTS AND METHODS Primary outcome 1.Is to assess the efficacy using stone free rate defined as no or stone fragment residual ≤ 4 mm by non-contrast computed tomography (NCCT) 3 months after the procedure.

Secondary outcomes

1.To assess the operative time, fluoroscopy time, haemoglobin drop, hospital stay, retreatment rate, ancillary procedure and the complications using the Clavien-Dindo system as described at European Association of Urology Guidelines Panel in Reporting and grading of complications after urologic surgical procedures.

Study Design:

The design of the research will be a prospective randomised controlled study. Study Setting/Location The study will be conducted in a single tertiary centre at urology department at Ain Shams University Hospital, Egypt.

Parents of eligible children presented with renal stone will be asked to participate in this study and will be provided with an informed consent form in line with Good Clinical Practise and the Declaration of Helsinki.

I.Eligibility Criteria

Inclusion criteria are:

1. Children from ages 2 to 12
2. Single renal stone pelvic, upper or middle calyceal
3. Stone diameter between 1 and 2 cm in the longest axis by NCCT
4. High-density (≥1000 HU) by NCCT

The exclusion criteria are:

1. Radiolucent stones
2. Co-existing renal anomalies
3. Acute UTI
4. Uncorrectable bleeding disorders
5. Musculoskeletal deformities
6. Patients with ureteral stones or ureteral obstruction Enrollment of the participants All patients will be assessed preoperatively by detailed medical history, physical examination, urinalysis, urine culture, kidneys, ureters and bladder (KUB) x-ray, renal ultrasonography (US) and a NCCT, as well as a routine preoperative evaluation.

Randomization and allocation Eligible and consenting participants will be randomized in 2 equal groups to intervention mini-PNL or SWL group. Randomization will be produced with a computer-generated program in permuted blocks of random lengths Technique All procedures will be done under general anesthesia.

1. Mini-PNL: All procedures will be done in the prone position. The target calyx will be punctured using fluoroscopic guidance with an 18-GA sheathed needle, and tract dilatation will be achieved using Amplatz dilators up to 16-18 Fr according to patient age. The holmium: YAG laser will be used to perform the stone fragmentation. Standard 12-Fr rigid nephroscope will be used for stone retrieval and fragmentation. A clamped nephrostomy tube will be placed routinely to reduce the bleeding for 24 h in all cases. The nephrostomy tube and the ureteral catheter will be removed on first and second postoperative days if there will be no complications.
2. SWL: The lithotripsy will be performed by an electromagnetic shockwave lithotripter (Dornier Compact Sigma). The lung and genitourinary fields will be shielded for all patients. Fluoroscopy will be used to localize the stone and to monitor fragmentation. The dispensed shockwave will begin at 14 kV and escalates to its maximum power level of 20 kV. The maximum number of shocks given per session will be between 1000 and 2500 depending on patient age (1000 waves per session for children younger than 5 years and 2500 waves per session for older children, with a frequency of 70 shocks/minute). The SWL session will be stopped when no visible stone is detected, or when tiny fragments are the only visible stone remnants, or when the desired number of shocks has been given.

Follow up:

Patients will be assessed 2 weeks after the procedure by KUB and US to assess SFR. SWL will be repeated in cases with residual stone fragments > 4mm for a maximum of 3 sessions. NCCT will be performed at 3 month post the procedure to assess the final SFR.

The following data will be recorded: patient age, gender, BMI, patient's complaint, stone location and diameter, operative and fluoroscopy time, hemoglobin drop, postoperative complications, hospital stay, need for retreatment, auxiliary procedures, and stone free rate.

STATISTICAL CONSIDERATIONS AND DATA ANALYSIS Sample size and statistical power Using G* power programme and chi-square test to calculate sample size. During the study, the minimal accepted total sample size will be 40 based on effect size of 0.76 based on the previous trial published recently (12) with a 99 % power "beta", 0.05 level of significance is considered "alpha". The sample size will be increased to be 40 patients in each group due to expected dropout rate.

Statistical Analysis Continuous data will be summarized using the mean ± SD and compared by t test. Categorical variables will be compared using the χ2 test or Fisher's exact test. The Statistical Package for Social Sciences, version 13.0, for Windows (SPSS, Chicago, IL) will be applied for statistical analysis. P≤.05 will be considered statistically significant.

Compliance with ethical standards Conflict of interest: The authors declare that they have no conflict of interest.

Human and animal rights: All procedures in this study involving human participants were in accordance with the 1964 Helsinki Declaration and its later amendments.

Informed consent: Informed consent will be obtained from all individual participants in this study

ELIGIBILITY:
Inclusion Criteria:

1. Children from ages 2 to 12
2. Single renal stone pelvic, upper or middle calyceal
3. Stone diameter between 1 and 2 cm in the longest axis by NCCT
4. High-density (≥1000 HU) by NCCT

Exclusion Criteria:

1. Radiolucent stones
2. Co-existing renal anomalies
3. Acute UTI
4. Uncorrectable bleeding disorders
5. Musculoskeletal deformities
6. Patients with ureteral stones or ureteral obstruction

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-05-28 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy assessed as stone free rate | 3 months
  defined as no or stone fragment residual ≤ 4 mm by non-contrast computed tomography (NCCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the IPD and supporting information will be available (1-feb-2026) and for how long (31-jun-2026).
Access Criteria: Who can access the IPD?
  * Any qualified researcher
  * Researchers with an approved proposal
  * Only collaborators or sponsors
  * Researchers affiliated with an academic institution
  What can they access?
  * De-identified individual participant data
  * Data underlying published results
  Supporting documents ( study protocol, statistical analysis plan, data dictionary)
  How can they access it?
  * By submitting a research proposal
  * After signing a data use or confidentiality agreement
  * Through a secure data-sharing platform or repository
  * By contacting the study sponsor or principal investigator